CLINICAL TRIAL: NCT06896175
Title: Effect of Ilex Paraguariensis Harvest Time and Consumption Method of Processed Yerba Mate on the Lipid Profile of Consumes in the Department of Caaguazu, Paraguay
Brief Title: Effect of Ilex Paraguariensis Harvest Time and Consumption Method of Processed Yerba Mate on the Lipid Profile
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Caaguazu (Other)
Collaborators: Hospital Nacional de Itaugua, MSPyBS, Paraguay) (Unknown); Instituto Nacional de Salud, Paraguay (Other); Universidad de La Frontera (Other); McMaster University (Other); Universidad del Cauca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PINV01-1074
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Lipid Metabolism Disorders
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: First, they will be divided into two groups: YMA (Yerba harvested at the beginning of the safra) and YMB (Yerba harvested at the end of the safra). Both groups are then divided into three strata: consumption of mate only, consumption of terere only, consumption of both mate and terere.
Who Masked: Participant, Care Provider, Investigator
Masking Description: They will not distinguished if the yerba is the harvested before or after the safra period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- YM mate (Active Comparator): Yerba consumption of mate only
  Interventions: Dietary Supplement: Yerba mate consumption (Ilex paraguayensis) A; Dietary Supplement: Yerba mate comsuption (ilex paraguayencis) B
- YM terere (Active Comparator): Yerba mate terere consumption only
  Interventions: Dietary Supplement: Yerba mate consumption (Ilex paraguayensis) A; Dietary Supplement: Yerba mate comsuption (ilex paraguayencis) B
- YM mate and terere (Experimental): Yerba mate consuptiom as mate and terere
  Interventions: Dietary Supplement: Yerba mate consumption (Ilex paraguayensis) A; Dietary Supplement: Yerba mate comsuption (ilex paraguayencis) B

INTERVENTIONS:
Dietary Supplement: Yerba mate consumption (Ilex paraguayensis) A — Yerba mate of the begining of the harvest time
Dietary Supplement: Yerba mate comsuption (ilex paraguayencis) B — Yerba mate of the final time of the harvest

SUMMARY:
Introduction: This project studies the impact of Ilex paraguariensis harvest time, commonly known as yerba mate, and its consumption mode (mate, tereré, and mate/terere) on the lipid profile of consumers in the Department of Caaguazú, Paraguay. Yerba mate is rich in bioactive compounds such as polyphenols, xanthines, and saponins. There are no clinical trials conducted in Paraguay with our Ilex paraguariensis plantations that have analyzed the influence of harvest time on the yerba mate production process and the infusion mode, in relation to its effect on dyslipidemias. General Objective: To establish the effectiveness of Ilex paraguariensis harvest time and the mode of consumption of the produced yerba mate on the lipid profile of consumers in the Department of Caaguazú, Paraguay. Methodology: The research approach will be quantitative, using a triple-blind randomized clinical trial design. Participants will be regular consumers of yerba mate, divided into groups based on harvest time (beginning or end of the harvest) and consumption mode (mate, tereré, or both). Lipid profile measurements will be taken at baseline and at 30, 90, and 180 days after consumption. Yerba mate samples will be analyzed and classified according to their bioactive properties before being blinded to the researchers and participants. Expected results: a report on the social, cultural, and anthropometric characterization of regular consumers of mate and tereré, and a report on the concentrations of the bioactive properties of yerba mate; polyphenols, xanthines, saponins from Ilex paraguariensis harvested at the beginning and end of the harvest and the database of patients with baseline lipid profile results, at 30, 90, and 180 days of mate and tereré consumers with yerba mate prepared randomly according to the harvest time of the Ip (beginning or end of harvest) analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals of both sexes, between 18 and 60 years of age, residing in the country, who consume prepared yerba mate.
2. Consumers of mate or tereré and mate/terere who agree to consume the yerba mate samples provided by the research team, which will be masked from laboratory analysis.
3. Two weeks of abstinence from consuming prepared yerba mate, either as mate or tereré, prior to randomization for the trial.
4. Consume exclusively prepared yerba mate in the prescribed manner (quantity of yerba, frequency of consumption, and sips), either in its mate or tereré form independently, and for those who consume both forms daily.
5. Do not change the yerba mate consumer's usual diet or regular physical activity during the trial period.
6. Agree to know the laboratory results of the lipid profile only at the end of the trial (180 days after the start).

Exclusion Criteria:

1. Individuals receiving lipid-lowering treatment at the start of the trial.
2. Consuming any other type of yerba mate not provided by the principal investigator.
3. Individuals requiring vitamins as a nutritional supplement.
4. Individuals taking thermogenic supplements.
5. Individuals consuming cooked mate.
6. Addiction to medicinal plants or herbs, both mate and tereré.
7. Individuals with a personal history of coronary artery disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 198 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Effect on lipid profile | six months
  Effect of total cholesterol, LDL, HDL and tryglicerids

CONTACTS AND LOCATIONS:
Overall Officials: Guiomar Viveros, Study Chair — Universidad Nacional de Caaguazu, Facultad de Ciencias de la Salud; Gloria Gonzalez, Study Director — Universidad Nacional de Caaguazu, Facultad de Ciencias de la Salud; Angel Rolon, Principal Investigator — Universidad Nacional de Caaguazu, Facultad de Ciencias de la Salud

IPD SHARING:
Plan to Share IPD: Undecided
It could be shared with anonimous data for the participants